CLINICAL TRIAL: NCT02948400
Title: Virtual Reality by Mobile Phone: Improving Child Pedestrian Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Drexel University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Schwebel, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD088415-01 (NIH); R01HD088415 (NIH)
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Child Pedestrian Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Google Cardboard virtual environment (Experimental): pedestrian safety training using the Google Cardboard device and delivery of a pedestrian virtual environment by mobile smartphone. Note that children in this arm will be trained using an immersive virtual environment delivered by smartphone, which is different from the other arm that is trained using a semi-immersive virtual environment delivered in a kiosk. The intervention is pedestrian safety training for both arms.
  Interventions: Behavioral: pedestrian safety training in pedestrian virtual environment
- semi-immersive virtual environment (Active Comparator): pedestrian safety training using a semi-immersive virtual pedestrian environment kiosk. Note that children in this arm will be trained using a semi-immersive virtual environment delivered in a kiosk, which is different from the other arm that is trained using an immersive virtual environment delivered by smartphone. The intervention is pedestrian safety training for both arms.
  Interventions: Behavioral: pedestrian safety training in pedestrian virtual environment

INTERVENTIONS:
Behavioral: pedestrian safety training in pedestrian virtual environment — pedestrian safety training

SUMMARY:
The investigators will conduct a non-inferiority clinical trial to evaluate whether children trained in pedestrian safety amidst a Google Cardboard virtual environment achieve equivalent levels of pedestrian safety to children trained in a full semi-immersive virtual pedestrian environment

ELIGIBILITY:
Inclusion Criteria:

* children ages 7-8 and their families
* one sibling per family, randomly chosen if multiple siblings are eligible
* children and parent speak English

Exclusion Criteria:

* disabilities that prohibit participants from valid understanding of or participation in the experimental protocol
* families that plan to move more than 50 miles away over the next year
* families unable to commit to frequent visits required in the study protocol

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
will share with qualified investigators upon their individual request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data available after all primary analyses are completed, for undetermined amount of time
Access Criteria: Data can be accessed by qualified investigators upon contacting the PI or study biostatitician

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were excluded prior to randomization, for the following reasons: COVID-related research closure: 2 Child discovered to be wrong age (ineligible): 5 Child unable to understand protocol: 1 Sibling discovered to be in study previously (ineligible): 3 Motion sickness in virtual reality: 1 Participant withdrew for unknown reasons: 9
Period: Overall Study
Arm/Group | Google Cardboard Virtual Environment | Semi-immersive Virtual Environment
Started | 254 | 225
Completed | 181 | 179
Not Completed | 73 | 46
Not completed — Withdrawal by Subject | 17 | 10
Not completed — failed to attend appointments | 47 | 34
Not completed — COVID-related closure | 6 | 2
Not completed — sibling discovered to be in study so participant ineligible | 1 | 0
Not completed — motion sickness in virtual reality | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Google Cardboard Virtual Environment | Semi-immersive Virtual Environment | Total
Number analyzed (Participants) | 254 | 225 | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (0.5) | 7.4 (0.5) | 7.5 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 118 | 257
  Male | 115 | 107 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 243 | 215 | 458
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 132 | 112 | 244
  White | 99 | 95 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 254 | 225 | 479

OUTCOME MEASURES:

1. Primary Outcome: Risky Crossings
Description: risky crossings in virtual environment setting, indicated by hits/close calls while crossing virtual street
Time Frame: 3.5 months after baseline (about 1 week after completion of all training)
Population: Participants who completed study protocol, as described in participant flow section
Measure: Mean (Standard Deviation); unit: count of risky crossings
Arm/Group | Google Cardboard Virtual Environment | Semi-immersive Virtual Environment
Number analyzed (Participants) | 181 | 179
count of risky crossings | .20 (.11) | .13 (.091)

ADVERSE EVENTS:
Time Frame: During participation in the study, about 6 months for each participant.
Description: The definition matches that in clinicaltrials.gov and requirements of our university IRB.
Arm/Group | Google Cardboard Virtual Environment | Semi-immersive Virtual Environment
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/225
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/225
Other Adverse Events (participants affected / at risk) | 1/254 | 0/225
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Google Cardboard Virtual Environment (N=254) | Semi-immersive Virtual Environment (N=225)
motion sickness (Nervous system disorders) | 1 (1) | 0 (0) — participant experienced possible fainting episode due to motion sickness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT02948400/Prot_SAP_000.pdf